CLINICAL TRIAL: NCT06262776
Title: Safety and Immunogenicity of Recombinant Zoster Vaccine for Kidney Transplant Recipients (SIR ZOSTER)
Brief Title: Safety and Immunogenicity of Recombinant Zoster Vaccine for Kidney Transplant Recipients
Acronym: SIR ZOSTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Adelaide Local Health Network Incorporated (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Adelaide (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Principal Investigator, Matthew Tunbridge, Principal Investigator, Central Adelaide Local Health Network Incorporated
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SIRZOSTER1.01
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Immunosuppression; Vaccine Response Impaired

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccination group (Experimental): All participants will receive the assigned intervention, a 2-dose course of Zoster recombinant adjuvanted vaccine. Study participants will include kidney transplant recipients receiving specific immunosuppressive medications, and non-immunosuppressed household cohabitants, with comparisons made in magnitude of vaccine response.
  Interventions: Biological: Recombinant zoster vaccine adjuvanted (SHINGRIX)

INTERVENTIONS:
Biological: Recombinant zoster vaccine adjuvanted (SHINGRIX) — 2 doses of 0.5mL recombinant zoster vaccine adjuvanted intramuscular injection at week 0 and week 8.

SUMMARY:
The goal of this clinical trial is to compare responses to Varicella Zoster vaccination between kidney transplant patients on different medication regimens, and their healthy co-habitants. The main questions it aims to answer are:

1. Are there differences in vaccination immunological responses in kidney transplant patients on different immunosuppression regimens?
2. Are there differences in vaccination immunological responses between kidney transplant patients and their healthy co-habitants? Participants will all receive a 2-dose course of SHINGRIX recombinant Zoster vaccination, and have immunological responses measured and compared at 5 timepoints between 1 week to 1 year post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Single organ kidney transplant recipient, currently receiving a specific immunosuppression regimen:

  1. Calcineurin inhibitor (tacrolimus or cyclosporine), antimetabolite (mycophenolate derivative or azathioprine), and oral steroid (n = 30)
  2. Calcineurin inhibitor (tacrolimus or cyclosporine), mTOR inhibitor (sirolimus or everolimus), and oral steroid (n = 30)
  3. mTOR inhibitor (sirolimus or everolimus), antimetabolite (mycophenolate derivative or azathioprine), and oral steroid (n = 30)
* Aged >18 years
* estimated glomerular filtration rate (GFR) > 15 mL/min/1.73m2
* Previous documented infection with Varicella zoster (known infection history or positive Varicella zoster IgG result)

OR

* Healthy household cohabitant of kidney transplant recipient enrolled in trial (n = 30)
* Aged > 50 years
* Previous documented infection with Varicella zoster (known infection history or positive Varicella zoster IgG result)

Exclusion Criteria:

* Unable or unwilling to provide informed consent to participate in the trial
* No previous infection with Varicella zoster (chickenpox)
* Known allergy to or intolerance of the contents of the SHINGRIX vaccine
* Current pregnancy
* For healthy household cohabitants, history of primary immunodeficiency, documented vaccine hypo-responsiveness, or active immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Functional T cell memory | 3 weeks following second vaccine dose
  ELISpot measurement of interferon gamma spot-forming units following 18-hour stimulation of peripheral blood mononuclear cells with Zoster gE protein-derived peptide array

SECONDARY OUTCOMES:
Frequency of virus specific T cells | 3 weeks and 52 weeks following second vaccine dose
  Change in frequency of CD8+ Zoster gE protein-specific T cells identified by flow cytometry as CD8+CD134+CD69+ following 24-hour stimulation with a gE protein-derived peptide array
Magnitude of antibody response | 3 weeks and 52 weeks following second vaccine dose
  Anti Varicella zoster gE Immunoglobulin M (IgM) and IgG antibody titres compared to baseline
Concentration of post-vaccination circulating cytokines | 3 weeks following second vaccine dose
  Post-vaccination circulating cytokines compared to baseline
Frequency of polyfunctional T cells | 3 weeks and 52 weeks following second vaccine dose
  Change in frequency of Zoster gE protein-specific polyfunctional T cells identified by flow cytometry intracellular cytokine staining (interferon-gamma, interleukin-2, tumour necrosis factor) following 24-hour stimulation with a gE protein-derived peptide array.
Magnitude of vaccine-induced cross-protective antiviral responses | 3 weeks and 52 weeks following second vaccine dose
  T cells will be investigated for cross-protective herpesviridae responses using interferon gamma ELISpot compared to baseline following 24-hour stimulation with a gE protein-derived peptide array.
Frequency of virus-specific T stem cell memory compared to baseline | 3 weeks and 52 weeks following second vaccine dose
  Frequency of Zoster gE protein-specific T stem cell memory (Tscm) will be determined by flow cytometry based on expression of T cell phenotypic markers (CD27+CD45RA+CD95+) on activation-induced marker-positive CD4 and CD8 T cells

OTHER OUTCOMES:
Incidence of shingles | 12 months
  Incidence of shingles in the study cohort from 3 weeks post-vaccination to 12 month follow-up
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  Safety of two-dose Zoster recombinant vaccine adjuvanted as measured by reported adverse events following immunisation using CTCAE v4.0 1 and 3 weeks after each vaccination, and 12 months after vaccination.
Tolerability of vaccination regimen as assessed by EQ-5D | 3 weeks following second vaccine dose
  Tolerability of two-dose Zoster recombinant vaccine adjuvanted as measured by quality of life questionnaire EuroQol-5 dimensional (EQ-5D) questionnaire at baseline and 3 weeks after second vaccine dose. This questionnaire assesses quality of life rated on a scale of 0 (worst) to 100 (best), and assesses functional capacity rated on a scale of 0 (best) to 5 (worst) across 5 domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Coates, FRACP, Principal Investigator — Central and Northern Adelaide Renal and Transplantation Services
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Identifiable data will not be publicly released, however, de-identified data will be made available in combination with publication of study results either as supplementary material or on public repository. Study protocol and statistical analysis plan will be made available as supplementary material with publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available following publication of trial results, and will be available in perpetuity.
Access Criteria: Trial results and supporting information outlined above will be made available through open access publishing.